CLINICAL TRIAL: NCT07000292
Title: A Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics and Efficacy of Subcutaneous Injection of MSC303 for the Treatment of Immune Glomerular Diseases
Brief Title: MSC303 Subcutaneous Injection for the Treatment of Immunologic Glomerular Disease.
Acronym: MSC303
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xu huji, Professor and Chief Physician, Head of the Department of Rheumatology and Immunology, Shanghai Changzheng Hospital., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC303-CT201
Record Dates: First submitted 2025-05-29; First posted 2025-06-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Lupus Nephritis (LN); ANCA-Associated Glomerulonephritis
Keywords: MSC303; Immune glomerular diseases
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC303 (Experimental): MSC303 is an asymmetric trivalent bispecific antibody targeting both CD20 and CD3 (with a ratio of CD20:CD3 at 2:1). By binding to the CD20 antigen on the surface of B cells with one end and the CD3 on the surface of T cells with the other, MSC303 recruits activated T cells around B cells, thereby enhancing the killing effect on B cells.
  Interventions: Drug: Injection of MSC303

INTERVENTIONS:
Drug: Injection of MSC303 — Dose Group 1: D1, D8, D15, and D36 were respectively given 1, 5, 15, and 15 mg of MSC303 for injection; The second dose group: D1, D8, D15 and D36 were respectively given for injection MSC303 1, 5, 20, 20 mg.

SUMMARY:
This study will evaluate the safety and efficacy of MSC303 in patients with Immune glomerular diseases.

DETAILED DESCRIPTION:
The primary endpoint of Phase Ib：Evaluate the safety of MSC303 in patients with Lupus Nephritis (LN）and ANCA-associated glomerulonephritis (ANCA-GN).

The primary endpoint of Phase II：Evaluate the change of Urine Protein/Creatinine Ratio (UPCR) in Week 12 compared with the baseline of MSC303 in patients with Lupus Nephritis(LN） and ANCA-associated glomerulonephritis (ANCA-GN).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years (including boundary values), gender unspecified；
2. Willing to participate voluntarily in this clinical study and with good compliance；
3. Regarding the criteria for the study diseases, meet the diagnostic criteria for any of the following diseases:

   1. Diagnosed with lupus nephritis(LN);
   2. diagnosed with ANCA-associated glomerulonephritis (ANCA-GN);
4. Sufficient organ function;

Exclusion Criteria:

1. History of severe allergic reaction to humanized monoclonal antibodies, or known allergy to any component of MSC303；
2. Active infection requiring antibiotic treatment；
3. Concomitant with other serious diseases；
4. Patients with congenital immunoglobulin deficiency；
5. Infection with human immunodeficiency virus (Human immunodeficiency virus (HIV)), hepatitis B or hepatitis C (including HBsAg, HBcAb positive with abnormal Hepatitis B Virus DNA (HBV DNA) or Hepatitis C virus RNA (HCV RNA ));
6. Other exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: safety Phase II: Urine Protein/Creatinine Ratio (UPCR) | 12 week
  Phase Ib: To evaluate the safety of MSC303 for injection in subjects with immune glomerular diseases.
  Phase II: To evaluate the change in Urine Protein/Creatinine Ratio (UPCR) from baseline at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Huji Xu, Ph.D, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding the security of patient personal information.